CLINICAL TRIAL: NCT06697444
Title: Risk Factors and Disorders Associated With Uterine Adenomyosis Diagnosed on Magnetic Resonance Imaging in Women of Reproductive Age
Brief Title: Risk Factors and Disorders Linked to Uterine Adenomyosis on MRI in Reproductive-Age Women
Status: Completed | Type: Observational
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Narges Afzali, Clinical Professor, Mashhad University of Medical Sciences
Other Study IDs: IR.IAU.MSHD.REC.1399.061
Record Dates: First submitted 2024-11-14; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Adenomyosis; Endometriosis; Leiomyoma (Uterine Fibroids); Ovarian Cysts
Keywords: Adenomyosis; magnetic resonance imaging; risk factors
MeSH Terms: conditions — Adenomyosis; Endometriosis; Leiomyoma; Ovarian Cysts

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational case-control study is to identify risk factors and associated conditions related to adenomyosis in women of reproductive age.

The main questions it aims to answer are:

Is there an association between a history of uterine surgery and the occurrence of adenomyosis? Does a higher prevalence of endometriosis or increased number of pregnancies correlate with adenomyosis? Researchers will compare women with MRI-confirmed adenomyosis to a control group of women who underwent pelvic MRI for other reasons but were not diagnosed with adenomyosis to see if there are significant differences in risk factors such as endometriosis, number of pregnancies, and history of uterine surgery.

Participants will:

Undergo pelvic MRI with and without intravenous contrast Provide information on factors such as age, smoking, number of pregnancies, history of uterine surgery, and coexisting conditions like leiomyoma and ovarian cysts This study aims to inform better management strategies for reducing the incidence of adenomyosis by targeting modifiable risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age (18-50 years).
* Patients who underwent pelvic MRI for clinical indications.
* MRI-confirmed diagnosis of adenomyosis (for the case group).
* Patients without adenomyosis confirmed by MRI (for the control group).
* Willingness to participate and provide informed consent.

Exclusion Criteria:

* Women outside the reproductive age range (under 18 or over 50 years).
* Pregnancy or lactation at the time of MRI.
* Previous hysterectomy or other major uterine surgeries.
* Presence of malignancies or other serious conditions that could interfere with the study.
* Inability to undergo MRI due to contraindications (e.g., metal implants, pacemakers).
* Incomplete or missing MRI data.
* Non-consent to participate in the study.

Max Age: 50 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes — Only individuals who self-identify as female were eligible to participate in this study, as it focused on conditions specific to the uterus.
Study Population: Case Group: 50 women of reproductive age (18-50 years) who were diagnosed with adenomyosis based on MRI findings.
  Control Group: 50 women of reproductive age (18-50 years) who underwent pelvic MRI for various clinical reasons but were not diagnosed with adenomyosis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of Endometriosis in Participants Diagnosed with MRI-Confirmed Adenomyosis | From admission to discharge, up to 1 week
  he presence of endometriosis will be evaluated in participants who have been diagnosed with adenomyosis through pelvic MRI. Diagnosis will be confirmed based on established imaging criteria, including areas of low signal intensity on T2-weighted MRI images. The prevalence will be compared between the case group (women with adenomyosis) and the control group (women without adenomyosis). The outcome will be reported as the percentage of participants in each group diagnosed with endometriosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Mashhad Medical Sciences, Islamic Azad University, Mashhad, Iran

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT06697444/SAP_000.pdf